CLINICAL TRIAL: NCT06644716
Title: [18F]F-FAPI PET-CT to Identify Carcinoma of Unknown Primary Origin
Acronym: FAPI for CUP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Cancer Society (Other); Academisch Ziekenhuis Maastricht (Other); Missie Tumor Onbekend (Unknown); Noordwest Ziekenhuisgroep (Other); Cyclotron Noordwest BV (Unknown)
Responsible Party: Principal Investigator, Dr. S.E.M. Veldhuijzen van Zanten, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-505592-69-00
Record Dates: First submitted 2024-10-04; First posted 2024-10-16 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Cancer of Unknown Primary
Keywords: [18F]F-FAPI; PET-CT; Cancer of Unknown Primary; Diagnostics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with CUP (Experimental): Patients diagnosed with CUP after standard diagnostic work-up including an [18F]FDG PET-CT
  Interventions: Diagnostic Test: [18F]F-FAPI PET-CT

INTERVENTIONS:
Diagnostic Test: [18F]F-FAPI PET-CT — Each patient will receive a FAPI PET-CT.

SUMMARY:
The investigators will determine the proportion of CUP patients in whom the primary tumor can be identified by [18F]F-FAPI PET-CT.

DETAILED DESCRIPTION:
Carcinoma of unknown primary origin (CUP) is a diverse group of cancers defined by the presence of metastatic disease with no identified primary tumor after exhaustive diagnostic work-up. Absence of a known targetable primary tumor precludes patients from receiving tumor-specific evidence-based therapies which significantly impacts the life expectancy of CUP patients. In this investigator-initiated and patient association-driven, multi-center, prospective clinical study we aim to detect the primary tumor by PET-CT using the novel radiotracer [18F]F-fluoro fibroblast activation protein inhibitor (F-FAPI). We will include 50 patients (aged >18 year) who have been diagnosed with CUP after standard diagnostic work-up including FDG PET-CT. Participation in the study entails a one-time [18F]F-FAPI PET-CT examination in one of the six study centers (UMC Groningen, UMC Utrecht, Antoni van Leeuwenhoek, Radboudumc, Maastricht UMC, Erasmus MC). For the interpretation of images, central reading will be performed and results will be made available to the treating physician with an accompanying recommendation for additional diagnostics and/or treatment. After 6 months, the results of the [18F]F-FAPI PET-CT will be compared with patient follow up, including clinical, radiological and pathological outcome parameters. These findings will holistically be discussed in a multidisciplinary Truth Panel meeting to determine a uniform verdict with regard to the clinical value of [18F]F-FAPI for CUP. We hypothesize that [18F]F-FAPI PET-CT will detect the primary tumor in at least 15% of our CUP patients.¬

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Histologically-confirmed metastatic disease without identification of a primary tumor after standard diagnostic work-up, according to the national care pathway for CUP (in Dutch: Regionaal Zorgpad Primaire Tumor Onbekend), which includes at least an [18F]FDG PET-CT.

Exclusion Criteria:

* Patients with metastasis from a known primary tumor.
* Sarcomas, melanomas, germ cell tumors, neuroendocrine tumors and haematological malignancies whose exact site of origin is not established.
* History of malignancy within 5 years prior to [18F]F-FAPI PET-CT scan, with the exception of the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in-situ of the cervix, nonmelanoma skin carcinoma, localized prostate cancer, ductal carcinoma in-situ, or Stage I uterine cancer.
* Prior systemic therapy for the treatment of CUP.
* Radiotherapy prior to [18F]F-FAPI PET-CT. Off note: radiotherapy with palliative intent for symptomatic skeleton lesions is allowed.
* Impaired renal function, defined as eGFR (MDRD) <25 ml/min/1,73 m2. An exception can be made in consultation with the treating physician.
* WHO performance status >2 (Vademecum).
* Pregnancy/breastfeeding. For the latter, temporary discontinuation may be considered.
* Known allergic reaction to therapeutic radiopharmaceuticals
* Inability to lie still on the back for the duration of PET-CT
* Any (other) condition, disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that may affect the interpretation of the results, or which might contribute substantially to the patient's experience of study burden (such as non-suppressible claustrophobia)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Detection of the primary tumor by [18F]F-FAPI PET-CT | 2 years
  The proportion of CUP patients in whom the primary tumor can be identified by [18F]F-FAPI PET-CT

SECONDARY OUTCOMES:
Sensitivity, specificity, positive- and negative predictive value of [18F]F-FAPI PET-CT | 2 years
  These numbers will be calculated based on correlation between the outcome of the FAPI reading and the clinical outcome for the patient, i.e., correct or incorrect identification of a primary tumor (or not) by additional diagnostics or follow-up determined as such by a dedicated Truth Panel established for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Veldhuijzen van Zanten, Principal Investigator — Erasmus Medical Center
Locations (6):
- Netherlands (6):
  - Antoni van Leeuwenhoekziekenhuis, Amsterdam
  - UMC Groningen, Groningen
  - Maastricht UMC, Maastricht
  - Radboud UMC, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years after publication of the main results.
Access Criteria: Investigators who provide a sound proposal which has been approved by a review committee.
URL: https://research.weill.cornell.edu/sites/default/files/clinicaltrials.gov_data_sharing_plan_info_sheet_v1.0_01.04.2019.pdf